CLINICAL TRIAL: NCT01952769
Title: A Phase I/ II Clinical Trial of MDV9300 (Pidilizumab) in Diffuse Intrinsic Pontine Glioma
Brief Title: Anti PD1 Antibody in Diffuse Intrinsic Pontine Glioma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: antiPD1brainad2- HMO-CTIL
Record Dates: First submitted 2013-09-15; First posted 2013-09-30 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2015-10

CONDITIONS: DIPG
Keywords: anti PD1,diffuse pontine glioma
MeSH Terms: interventions — pidilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment of DIPG with MDV9300 (Experimental): treatment of diffuse pontine glioma with MDV9300 with the combination of radiation and low dose cyclophosphamide
  Interventions: Biological: MDV9300

INTERVENTIONS:
Biological: MDV9300 — The study will be done in the following manner:
  1. Evaluation of MDV9300 and radiation-
     1. Cohort A-3 patients: first dose of MDV9300 3mg/m2 .If no toxicity over grade 2-second dose and on -6 mg/kg.
     2. Cohort B -3 patiens: if no toxicity >grade 2 seen in cohort A- start dose will be 6 mg/kg If toxicity> grade 2 in 2 patients or more on a dose of 3 mg/kg the dose in cohort B will be 1 mg/kg during irradiation If toxicity> grade 2 in 2 patients or more on a dose of 1 mg/kg no further concurrent MDV9300 and radiation will be given
  2. Evaluation of MDV9300 and cyclophosphamide
  After completion of the first phase (6 patients) a cohort of 15 patients will be accrued. The treatment protocol of this cohort will be as follows:
  Following radiation completion , and after recovery from treatment adverse events of grade 2 and higher, the patients will be started on concurrent biweekly MDV9300 and weekly cyclophosphamide 200mg/m2
  Other Names: pidilizumab

SUMMARY:
Diffuse pontine gliomas are incurable with currently used treatments. based on data stating that progressive tumors inhibit immune system, would try to enhance immune system activity and tumor cell killing. anti PD1 prevents one of the important mechanisms allowing the tumor to supress the immune system thus we hope it will allow for prolonged control of the tumors

DETAILED DESCRIPTION:
1. Diffuse intrinsic pontine glioma Diffuse intrinsic pontine glioma (DIPG) is the most lethal pediatric malignant disease. Children are usually diagnosed at the age of 6-8 years following a short history of neurological deterioration with often a combination of cranial nerve dysfunction, ataxia and long tract deficits. Diagnosis is MRI based and a biopsy is required only when tumor features on imaging are non-classic . As of today there is no curative treatment regardless of multiple clinical trials done in the past. Following diagnosis children undergo radiation therapy aiming at symptoms alleviation, with almost inevitable disease progression taking place several months later. Overall survival ranges between 9-12 months and death due to disease progression is the rule (1)
2. Relapsed high grade glioma- closed to accrual
3. Immunotherapy in brain tumors Data regarding possible role of the immune system in cancer was first presented in 2001 when Schreiber and Old demonstrated that lymphocytes, activated by interferon-γ, inhibit the development of spontaneous and carcinogen-induced tumors in immunodeficient mice (Shankaran et al, 2001). Later studies demonstrated progressively decreasing immunogenicity in tumor cells of advanced cancer patients. Based on these and other data trials incorporating immunotherapy into treatment of relapsed high grade glioma were constructed. Past trials centered upon active cell based immunization trying to present the patients' immune system with specific antigens derived from their tumor while using different techniques to enhance immune response. These studies has shown positive results but the need to prepare patient specific vaccination limited their use to highly specialized centers and results were hard to reproduce.(3)
4. The role of PD-1 in cancer immunotherapy One of the mechanisms through which tumor cells escape immune detection is activation of the inhibitory lymphocyte receptor PD-1 (programmed death 1). Low grade activation of the T cell receptor-secondary to prolonged antigen exposure (as found in chronic disease or protracted exposure to malignant cells) - strongly activates- PD-1. Upon activation, PD-1 drives the lymphocyte towards apoptosis and reduces cytokine production. PD-1/PD-1 ligand interaction promotes tolerance of the immune system to a specific antigen (4). Lately, studies reported high levels of PD-1 expression in tumor infiltrating lymphocytes ,and strong expression of PD-ligand within multiple tumor types including high grade glioma .Both these findings support the data regarding the role of PD1 in cancer immune escape (5).
5. Anti PD-1:Safety and efficacy in human studies Over the last two years data has been accumulating regarding efficacy and toxicity profile of anti PD-1.Topalian et.al reported at 2012 outcome of a large phase I study evaluating antiPD-1 in advanced cancers. Out of 296 participating patients 14% had Grade 3 or 4 drug-related adverse events with most being treated on an outpatient setup . Several patients were diagnosed with pneumonitis. Most were observed or treated successfully with steroids but three patients died. Among 236 patients in whom response could be evaluated, objective responses (complete or partial responses) were observed in those with non-small-cell lung cancer-a cancer not known to be immunoresponsive (18%), melanoma (28% ), or renal-cell cancer (27%). Responses were durable; 20 of 31 responses lasted 1 year or more (6). Further studies report a better toxicity profile with similar efficacy. Hamid et.al reported outcome of 135 patients with advanced melanoma. Side effects were mostly grade 1-2 with no treatment related mortality. Response rate among these patients was 38% and most responses lasted at least 7 months (7). A study evaluating anti PD-1 in chronic HCV patient revealed similar safe profile. One patient out of 66 (10 mg/kg) experienced an asymptomatic grade 4 ALT elevation coincident with the onset of a 4-log viral load reduction. Six patients exhibited immune-related adverse events of mild-to-moderate intensity, including two cases of hyperthyroidism consistent with autoimmune thyroiditis (8).
6. Anti CTLA-4 and anti PD-1 activity in brain tumors Unlike chemotherapy or targeted therapies, both antiCTLA-4 and anti PD-1 affect T lymphocytes rather than the tumor itself. Binding to the lymphocyte receptor may take place outside of the central nervous system. Following binding to their receptor the reactivated lymphocytes penetrate the brain and arrive to the tumor thus the antibodies are not required to cross the blood brain barrier. Data regarding activity of antiCTLA-4 within the brain may be retrieved from retrospective summary of melanoma patients with brain metastasis. These patients are usually ineligible for clinical trials due to their grim prognosis. Margolin e al reported partial response in 5 patients and stable disease for 12 weeks in another 4 out of 51 patients with asymptomatic brain melanoma metastasis. Patients with symptomatic lesions requiring steroid therapy did not respond. Di Giacomo reported disease stabilization in 5 and near total response in another 5 patients out of 20 patients with asymptomatic metastatic melanoma lesions. These data provide proof of principle to the assumption that this regimen is active within the brain.

   Zeng et al reported improved survival of glioblastoma implanted mice following radiation and anti PD-1. Median survival was 25 days in the control arm, 27 days in the anti-PD-1 antibody arm, 28 days in the radiation arm, and 53 days in the radiation plus anti-PD-1 therapy arm, these data along with tolerability of treatment calls for a clinical trial assessing this treatment in this population with extremely poor prognosis (9).
7. MDV9300 mechanism of action and early efficacy data

MDV9300 is one of several humanized anti PD1 antibodies currently under investigation in multiple tumors. A single dose of MDV9300 given to mice with metastatic melanoma, fibrosarcoma, lung carcinoma or colorectal adenocarcinoma led to significant reduction in lung and/or liver metastases along with prolonged survival. Combination of MDV9300 with rituximab, chemotherapy and different types of vaccines has proven to be synergistic.

In a phase I study enrolling 17 patients with advanced stage hematological malignancies (AML,CLL, Non-Hodgkin lymphoma, Hodgkin's disease and multiple myeloma) 5 patients had prolonged stable disease (averaging 60 weeks) and one patient with follicular lymphoma had a complete response.

A Phase II study was conducted in 72 adult patients with DLBCL following autologous stem cell transplantation; in this study, MDV9300 was given at a dose of 1.5 mg/kg per patient at 3 cycles per patient every 42 days (treatment Days 1, 43, and 85). The PFS and OS 18 months after transplant were 72% and 85%, respectively. These values compare favorably with results obtained in previous similar cohorts. In addition, the ORR within the 40 patients who enrolled in the study with measurable disease was 45% (30%CR, 15%PR).

A Phase II study was conducted in 30 adult patients with rituximab-sensitive, grade 1-2 follicular lymphoma who relapsed after 1-4 prior therapies with measurable disease. MDV9300 was administered at 3 mg/kg IV every 4 weeks for 12 infusions and rituximab was dosed at 375 mg/m2 IV weekly for 4 weeks starting 2 weeks after the first infusion of MDV9300. Of the 29 patients eligible for efficacy analysis, 19 had an objective response for an ORR of 66%. CR was observed in 15 (52%) and PR in 4 (14%). Altogether, 25 (86%) patients had measurable tumor regression. The ORR of 66% and CR rate of 52% compare favorably with the previously reported ORR of 40% and CR rate of 11% with single agent rituximab retreatment in relapsed follicular lymphoma. Median time to response was 88 days. Of note, 17% of the patients achieved initial response >3 months from first treatment. Median PFS was 19.6 months, and was not reached for the 19 responders or the 25 patients with measurable tumor regression.

H. in the first part of this study eight patients were enrolled . A total of 73 cycles of MDV9300 (range 2- 16) were applied. Treatment was well tolerated, with a mild to moderate fatigue experienced by 10% of the patients following treatment (7 cycles). Nine cycles were followed by neutropenia (CTCEA grade 1-3). No patient was diagnosed with neutropenia of less than 500 cells /mm3. The only other grade 3 adverse event was a single event of transient blood pressure during MDV9300 infusion. Median overall survival was 13 months (6-19 months) with 50% survival at 1 year.

CONCLUSION: Anti PD1 treatment is a well-tolerated therapy with possible activity in DIPG.

ELIGIBILITY:
Inclusion criteria:

1. Age: 3-21
2. Diagnosis:

   a. DIPG diagnosed based on all the following: i. Symptoms starting less than 6 weeks prior to diagnosis ii. Symptoms include one or more of the following: cranial nerve deficit, cerebellar or long tract dysfunction iii. MRI reveals a lesion infiltrating>70% of the pons
3. patient status:

   1. karnofsky or lansky (for children) scale of 60 or more (see appendix I)
   2. liver function:Total bilirubin ≤ 2 ULN, ALT or AST ≤ 2.5 ULN (or < 5 in case of liver impairment)
   3. neutrophils ≥ 1,ooo/mm3, platelets ≥ 100,000/mm3,Lymphocytes ≥1000
   4. Serum creatinine ≤ 1.5 ULN
4. Life expectancy of at least 4 months
5. Pregnancy:

   1. Negative pregnancy test in women of childbearing potential
   2. Use of an effective contraceptive method during the whole treatment and up to 3 months after the completion of treatment in males and females
6. prior informed consent signed

Exclusion criteria:

1. Severe bacterial, viral or fungal infection (Grade > 2 NCI-CTCAE v.4.0)
2. Any other serious uncontrolled medical condition (including active bleeding or non healing wound)
3. Pregnant or breastfeeding women
4. Participation in another clinical trial up to 10 days prior to study entry
5. Steroid treatment in a dose more than to 3mg dexamethasone / m2 *
6. Past infection with HCV

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-11 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
treatment related toxicity | monthly for 1 year or if treatment will be continued further due to response-throughout treatment
  Treatment related toxicity according to NCI CTC Version 4.0 will be recorded throughout treatment. a patient with grade 3 or more treatment related toxicity will receive 50% dose reduction. if again grade 3 treatment related toxicity will occur the patient will be taken off study.

SECONDARY OUTCOMES:
progression free survival | 6 months
  tumor measurements according to RANO criteria will be recorded

OTHER OUTCOMES:
overall survival | 6 months
  survival after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Hospital, Jerusalem, Israel